CLINICAL TRIAL: NCT00413309
Title: Gastrointestinal Ulceration in Patients on Dual Antiplatelet Therapy After Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Samuel Z. Goldhaber, MD, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000376
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Antiplatelet Therapy; PillCam; Endoscopy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Videotape Recording; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Video Capsule Endoscopy — Noninvasive pill endoscopy is undertaken after 90 days of Aspirin/Clopidogrel in patients who have had percutaneous coronary intervention with drug-eluting stents.
  Other Names: PillCam

SUMMARY:
To determine the rate of symptomatic and asymptomatic gastrointestinal erosions and ulcerations in patients on dual antiplatelet (aspirin and clopidogrel) therapy after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Background and Significance:

Percutaneous coronary intervention (PCI) is the standard of care for patients with acute coronary syndrome (ACS). Approximately 1,200,000 PCIs were performed in 2002 in the United States. Drug-eluting coronary stents have nearly abolished the clinical problem of in-stent restenosis at a cost of increased susceptibility to in-stent thrombosis, a catastrophic event associated with a 6-month mortality rate of 8.9% and a myocardial infarction rate that exceeds 50%.

To prevent in-stent thrombosis, PCI patients receive aspirin 325 mg and a minimum loading dose of clopidogrel 300 mg prior to stent deployment. In actual practice, many patients are now receiving a clopidogrel loading dose of 600 mg to ensure adequate platelet inhibition. Muller et al showed that administration of a higher loading dose (600mg) of clopidogrel to patients undergoing PCI accelerates suppression of platelet aggregation when evaluated by aggregometry. When patients were given a higher loading dose (600mg) of clopidogrel as opposed to the conventional loading dose (300mg), there was a 50% reduction in myocardial infarction after PCI in patients who received the higher dose. If a 600 mg loading dose of clopidogrel is adopted as routine practice, there may be a further increase in the risk of major gastrointestinal (GI) ulceration.

In multivariable analysis, the strongest predictor of stent thrombosis is premature discontinuation of dual antiplatelet therapy, exceeding other independent predictors such as renal failure, bifurcation lesions, diabetes, and low ejection fraction. Hence, following PCI with drug-eluting stents, dual antiplatelet therapy, with aspirin 75 to 162 mg lifelong in combination with clopidogrel 75 mg for at least 3 months, is prescribed.

The risk of overt GI bleeding with dual antiplatelet therapy can be as high as 1.3% within the first 30 days of therapy. Weil et al found that all doses of aspirin were associated with an increased risk of GI bleeding and that the risk of GI bleeding due to low-dose aspirin was dose-related: odds ratio 2.3 for 75 mg ⁄day; 3.2 for 150 mg ⁄day; 3.9 for 300 mg ⁄day. In the Clopidogrel for Unstable angina to prevent Recurrent Events (CURE) study, Peters et al showed that the risk of bleeding at the highest dose of aspirin (≥ 200mg) given with placebo was higher (3.7 %) than the risk of GI bleeding with the combination of clopidogrel and aspirin in the lowest dose group (3.0 %).

Kelly et al showed that the relative risks of upper GI bleeding for plain, enteric-coated, and buffered aspirin at average daily doses of 325 mg or less were 2.6, 2.7, and 3.1, respectively. Conventional thinking is that compared with the stomach, the relatively alkaline duodenum is less susceptible to aspirin-induced damage. However, Kelly et al found in contrast to conventional thinking that the relative risk point estimates for all three forms of aspirin were approximately the same for gastric and duodenal bleeding. A possible explanation is that systemic effects (e.g., on platelets and prostaglandin synthesis) are unlikely to differ according to the aspirin preparation used and may overwhelm any differences in local effects on the gastric or duodenal mucosa.

In addition to local irritation of the gastric mucosa, aspirin and other antiplatelet agents cause gastric damage through inhibition of prostaglandin synthesis and by producing microcirculatory injury. Antiplatelet drugs might interfere with gastric ulcer healing by suppressing the release of growth factors, such as vascular endothelial growth factor (VEGF), from platelets.

Patients who are at highest risk for GI bleeding while on antiplatelet therapy are the elderly, patients with history of gastric ulcers, gastroesophageal reflux disease (GERD), esophagitis, untreated Helicobacter pylori infection, intestinal polyps, cancer, and those with concomitant use of anticoagulants, steroids, or nonsteroidal anti-inflammatory drugs (NSAIDS). Patients on dual antiplatelet therapy can develop both upper and lower GI bleeding. GI hemorrhage is associated with an increased mortality rate, a greater need for surgery, blood transfusions, a prolonged length of hospital stay, and increased overall health care costs. While upper GI bleeding can be prevented with appropriate prophylaxis, there is no prophylaxis for lower GI bleeding.

Acid-suppressive therapy is beneficial in the prevention of upper GI bleeding. Two major classes of agents for the prevention of upper GI bleeding due to ulcer complications from antiplatelet therapy are: 1) acid-suppressive therapy with H2-antagonists and 2) proton pump inhibitors (PPIs). H2-antagonists exert their therapeutic effects by reversibly blocking H2-receptors on the basolateral membrane of gastric parietal cells. Until the early 1990s, H2-antagonists were the mainstay of pharmacotherapy for the prevention and management of upper GI bleeding. Between 1984 and 2000, 32 randomized controlled trials were conducted comparing H2-antagonists with placebo. Agents evaluated in these studies included cimetidine, ranitidine, and famotidine. Many were limited by small sample size and wide variations in study design. In a meta analysis of 11 randomized controlled trials with H2-antagonists, Koch et al showed that H2-antagonists did not prevent gastric ulcers, either in the short-term (< 2weeks) or long-term (>4weeks) of NSAID treatment. The average baseline risks for gastric ulcers were found to be 3.6% and 6.8% with short- and long-term NSAID treatment, respectively. The average baseline risks for gastric lesions were 53% and 27% with short- and long-term NSAID treatment, respectively. The H2 blockers did not lead to a significant risk reduction in gastric lesions during either short-term or long-term therapy. A statistical advantage of H2 blockers was shown only in 1 of 9 studies.

The average baseline risks for a duodenal ulcer were found to be 3% and 4% with short- and long-term NSAID treatment, respectively. The H2 blockers did not lead to a significant reduction in risk for duodenal ulcer during short-term treatment. A statistical advantage of H2 blockers was shown in 3 of 5 long-term studies, but in none of the 4 short-term trials. The average baseline risks for duodenal lesions were found to be 11% and 12% with short- and long-term NSAID treatment, respectively. The H2 blockers did not lead to a significant reduction in the risk for duodenal lesions, either during short-term or long-term treatment.

Factors limiting the utility of H2-antagonists include the development of tachyphylaxis, the need for dosage adjustment in renal insufficiency, thrombocytopenia, and mental status changes seen with higher doses of these medications. With the introduction of safer and more effective agents like PPIs, the role of H2-antagonists in the prevention and management of upper GI bleeding has diminished.

PPIs work by irreversibly inhibiting H+ pumps in gastric parietal cells. PPIs have a number of theoretical advantages over H2-antagonists. First, PPIs block the final step of acid production, negating stimulation of gastric secretion by gastrin, histamine, and acetylcholine, leading to prolonged acid suppression. Second, unlike H2-antagonists, tachyphylaxis has not been noted with PPIs.

Yeomans et al showed that omeprazole (PPIs) is more effective than H2 receptor antagonists in gastric acid suppression, preventing ulcers, and healing ulcers related to chronic use of NSAIDS.

In a randomized, open-label, five-way crossover study, the 24-h intragastric pH profile of oral esomeprazole 40 mg, lansoprazole 30 mg, omeprazole 20 mg, pantoprazole 40 mg, and rabeprazole 20 mg once daily in 34 patients with symptoms of gastroesophageal reflux disease was evaluated. Intragastric pH was maintained above 4.0 for a mean of 14.0 h with esomeprazole, 12.1 h with rabeprazole, 11.8 h with omeprazole, 11.5 h with lansoprazole, and 10.1 h with pantoprazole.

Esomeprazole also provided a significantly higher percentage of patients with an intragastric pH greater than 4.0 for more than 12 h relative to the other proton pump inhibitors. The frequency of adverse events was similar among treatment groups. Esomeprazole at the standard dose of 40 mg once daily provided more effective control of gastric acid at steady state than standard doses of other PPIs.

Chan et al randomized 320 patients with previous bleeding on aspirin to clopidogrel and placebo versus aspirin and esomeprazole. The cumulative incidence of ulcer bleeding in this study was 8.6% in patients who received clopidogrel and 0.7% in patients who received aspirin and esomeprazole.

Esomeprazole 40 mg once a day was found to be more efficacious than esomeprazole 20 mg once a day and 10 mg once a day in healing of erosive esophagitis and gastritis without significant difference in long-term safety or tolerability.

Esomeprazole is extensively metabolized in the liver by CYP3A4 but no clinically relevant interactions with drugs metabolized by the CYP system have been reported.

Assessment of GI Ulceration:

To detect GI ulcerations, endoscopy is the "gold standard". However, the invasiveness of traditional endoscopy in PCI patients with coronary artery disease makes this approach inappropriate.

An alternative imaging test that is noninvasive and does not require sedation is the PillCamÒ ESO capsule endoscope. The disposable, ingestible PillCamÒESO endoscope is an 11 X 26 mm capsule and acquires video images from both ends of the device during passage through the esophagus. The capsule transmits the acquired images via digital radiofrequency communication channel to the data recorder unit located outside the body.

The data recorder, an external receiving/recording unit is worn on patient's belt. It receives the data transmitted by the capsule. Upon completion of the examination, the physician transfers accumulated data in the data recorder is transferred to computer software for processing and interpretation.

The sensitivity of the PillCamÒ ESO in diagnosing any esophageal abnormalities is 92% and the negative predictive value (NPV) is 88%. Specificity and positive predictive value in diagnosing any esophageal abnormalities (PPV) are 95% and 97%, respectively.

The PillCamÒ ESO capsule is intended for visualization of the esophagus and not the stomach in adult patients, but detection of gastritis is feasible.

The PillCamÒ ESO capsule is contraindicated for use under the following conditions:

* Known or suspected GI obstruction, strictures, or fistulas based on the clinical picture or pre-procedure testing and profile.
* Cardiac pacemakers or other implanted electromedical devices.
* Swallowing disorders.

In this investigator-initiated trial, we will enroll 30 patients requiring dual antiplatelet therapy after PCI to determine the rate of occult and overt GI ulceration in patients on antiplatelet therapy after PCI. All patients will receive PillCamÒ ESO endoscopy after 80-90 days of aspirin and clopidogrel therapy to detect gastric erosions and ulcers. This will provide us with an event rate of GI ulceration in patients on dual antiplatelet therapy without acid suppressive medication prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone PCI within the preceding 72 hrs
2. Patients on aspirin and clopidogrel
3. Age greater than 18 years and less than 80 years
4. Written informed consent

Exclusion Criteria:

1. Active bleeding
2. Pregnancy
3. Patients already on H2 antagonists
4. Patients already on PPI
5. Patients with implanted cardiac defibrillator (ICD)
6. Patients with GI strictures, swallowing disorders, or bowel obstruction and fistulas.
7. Patients with significant gastrointestinal diverticular disease
8. Patients likely to require MRI imaging during the time the PillCam is still in the digestive tract (8 to 72 hours after the PillCam procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
A composite of overt and occult GI bleeding, gastritis, and esophageal, gastric, or duodenal ulcerations. | 90 Days
Overt GI symptoms include GI bleeding requiring hospitalization, blood transfusion, and/or interventions like endoscopy or surgery or gastroesophageal acid reflux (GERD) requiring acid-suppressive therapy. | 90 Days
Occult GI ulcerations and erosions include those detected by capsule endoscopy (PillCamÒ ESO) within 80 to 90 days after initiation of dual antiplatelet therapy. | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Smith SC Jr, Dove JT, Jacobs AK, Kennedy JW, Kereiakes D, Kern MJ, Kuntz RE, Popma JJ, Schaff HV, Williams DO, Gibbons RJ, Alpert JP, Eagle KA, Faxon DP, Fuster V, Gardner TJ, Gregoratos G, Russell RO, Smith SC Jr; American College of Cardiology/American Heart Association task force on practice guidelines (Committee to revise the 1993 guidelines for percutaneous transluminal coronary angioplasty); Society for Cardiac Angiography and Interventions. ACC/AHA guidelines for percutaneous coronary intervention (revision of the 1993 PTCA guidelines)-executive summary: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee to revise the 1993 guidelines for percutaneous transluminal coronary angioplasty) endorsed by the Society for Cardiac Angiography and Interventions. Circulation. 2001 Jun 19;103(24):3019-41. doi: 10.1161/01.cir.103.24.3019. No abstract available. PMID 11413094
- [Background] Patti G, Colonna G, Pasceri V, Pepe LL, Montinaro A, Di Sciascio G. Randomized trial of high loading dose of clopidogrel for reduction of periprocedural myocardial infarction in patients undergoing coronary intervention: results from the ARMYDA-2 (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2005 Apr 26;111(16):2099-106. doi: 10.1161/01.CIR.0000161383.06692.D4. Epub 2005 Mar 6. PMID 15750189
- [Background] Kastrati A, von Beckerath N, Joost A, Pogatsa-Murray G, Gorchakova O, Schomig A. Loading with 600 mg clopidogrel in patients with coronary artery disease with and without chronic clopidogrel therapy. Circulation. 2004 Oct 5;110(14):1916-9. doi: 10.1161/01.CIR.0000137972.74120.12. Epub 2004 Jul 19. PMID 15262828
- [Background] Muller I, Seyfarth M, Rudiger S, Wolf B, Pogatsa-Murray G, Schomig A, Gawaz M. Effect of a high loading dose of clopidogrel on platelet function in patients undergoing coronary stent placement. Heart. 2001 Jan;85(1):92-3. doi: 10.1136/heart.85.1.92. No abstract available. PMID 11119474
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; Canadian Cardiovascular Society. ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Revise the 1999 Guidelines for the Management of Patients with Acute Myocardial Infarction). Circulation. 2004 Aug 31;110(9):e82-292. No abstract available. PMID 15339869
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Weil J, Colin-Jones D, Langman M, Lawson D, Logan R, Murphy M, Rawlins M, Vessey M, Wainwright P. Prophylactic aspirin and risk of peptic ulcer bleeding. BMJ. 1995 Apr 1;310(6983):827-30. doi: 10.1136/bmj.310.6983.827. PMID 7711618
- [Background] Peters RJ, Mehta SR, Fox KA, Zhao F, Lewis BS, Kopecky SL, Diaz R, Commerford PJ, Valentin V, Yusuf S; Clopidogrel in Unstable angina to prevent Recurrent Events (CURE) Trial Investigators. Effects of aspirin dose when used alone or in combination with clopidogrel in patients with acute coronary syndromes: observations from the Clopidogrel in Unstable angina to prevent Recurrent Events (CURE) study. Circulation. 2003 Oct 7;108(14):1682-7. doi: 10.1161/01.CIR.0000091201.39590.CB. Epub 2003 Sep 22. PMID 14504182
- [Background] Kelly JP, Kaufman DW, Jurgelon JM, Sheehan J, Koff RS, Shapiro S. Risk of aspirin-associated major upper-gastrointestinal bleeding with enteric-coated or buffered product. Lancet. 1996 Nov 23;348(9039):1413-6. doi: 10.1016/S0140-6736(96)01254-8. PMID 8937281
- [Background] Ma L, Elliott SN, Cirino G, Buret A, Ignarro LJ, Wallace JL. Platelets modulate gastric ulcer healing: role of endostatin and vascular endothelial growth factor release. Proc Natl Acad Sci U S A. 2001 May 22;98(11):6470-5. doi: 10.1073/pnas.111150798. Epub 2001 May 15. PMID 11353854
- [Background] Lau WC, Gurbel PA, Watkins PB, Neer CJ, Hopp AS, Carville DG, Guyer KE, Tait AR, Bates ER. Contribution of hepatic cytochrome P450 3A4 metabolic activity to the phenomenon of clopidogrel resistance. Circulation. 2004 Jan 20;109(2):166-71. doi: 10.1161/01.CIR.0000112378.09325.F9. Epub 2004 Jan 5. PMID 14707025
- [Background] Rivkin K, Lyakhovetskiy A. Treatment of nonvariceal upper gastrointestinal bleeding. Am J Health Syst Pharm. 2005 Jun 1;62(11):1159-70. doi: 10.1093/ajhp/62.11.1159. PMID 15914876
- [Background] Levine JE, Leontiadis GI, Sharma VK, Howden CW. Meta-analysis: the efficacy of intravenous H2-receptor antagonists in bleeding peptic ulcer. Aliment Pharmacol Ther. 2002 Jun;16(6):1137-42. doi: 10.1046/j.1365-2036.2002.01274.x. PMID 12030956
- [Background] Koch M, Dezi A, Ferrario F, Capurso I. Prevention of nonsteroidal anti-inflammatory drug-induced gastrointestinal mucosal injury. A meta-analysis of randomized controlled clinical trials. Arch Intern Med. 1996 Nov 11;156(20):2321-32. PMID 8911239
- [Background] Yeomans ND, Tulassay Z, Juhasz L, Racz I, Howard JM, van Rensburg CJ, Swannell AJ, Hawkey CJ. A comparison of omeprazole with ranitidine for ulcers associated with nonsteroidal antiinflammatory drugs. Acid Suppression Trial: Ranitidine versus Omeprazole for NSAID-associated Ulcer Treatment (ASTRONAUT) Study Group. N Engl J Med. 1998 Mar 12;338(11):719-26. doi: 10.1056/NEJM199803123381104. PMID 9494148
- [Background] Miner P Jr, Katz PO, Chen Y, Sostek M. Gastric acid control with esomeprazole, lansoprazole, omeprazole, pantoprazole, and rabeprazole: a five-way crossover study. Am J Gastroenterol. 2003 Dec;98(12):2616-20. doi: 10.1111/j.1572-0241.2003.08783.x. PMID 14687806
- [Background] Chan FK, Ching JY, Hung LC, Wong VW, Leung VK, Kung NN, Hui AJ, Wu JC, Leung WK, Lee VW, Lee KK, Lee YT, Lau JY, To KF, Chan HL, Chung SC, Sung JJ. Clopidogrel versus aspirin and esomeprazole to prevent recurrent ulcer bleeding. N Engl J Med. 2005 Jan 20;352(3):238-44. doi: 10.1056/NEJMoa042087. PMID 15659723
- [Background] Johnson DA, Benjamin SB, Vakil NB, Goldstein JL, Lamet M, Whipple J, Damico D, Hamelin B. Esomeprazole once daily for 6 months is effective therapy for maintaining healed erosive esophagitis and for controlling gastroesophageal reflux disease symptoms: a randomized, double-blind, placebo-controlled study of efficacy and safety. Am J Gastroenterol. 2001 Jan;96(1):27-34. doi: 10.1111/j.1572-0241.2001.03443.x. PMID 11197282
- [Background] Maton PN, Vakil NB, Levine JG, Hwang C, Skammer W, Lundborg P; Esomeprazole Study Investigators. Safety and efficacy of long term esomeprazole therapy in patients with healed erosive oesophagitis. Drug Saf. 2001;24(8):625-35. doi: 10.2165/00002018-200124080-00006. PMID 11480494
- [Background] Eliakim R, Sharma VK, Yassin K, Adler SN, Jacob H, Cave DR, Sachdev R, Mitty RD, Hartmann D, Schilling D, Riemann JF, Bar-Meir S, Bardan E, Fennerty B, Eisen G, Faigel D, Lewis BS, Fleischer DE. A prospective study of the diagnostic accuracy of PillCam ESO esophageal capsule endoscopy versus conventional upper endoscopy in patients with chronic gastroesophageal reflux diseases. J Clin Gastroenterol. 2005 Aug;39(7):572-8. doi: 10.1097/01.mcg.0000170764.29202.24. PMID 16000923
- See also: North American Thrombosis Forum — http://www.natfonline.org